CLINICAL TRIAL: NCT01507636
Title: Apraxia-specific Occupational Therapy in Patients With Multiple Sclerosis
Brief Title: Occupational Therapy in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr. med. Christian Philipp Kamm, Department of neurology, University hopsital Bern, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 042/11
Record Dates: First submitted 2012-01-04; First posted 2012-01-11 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Sclerosis; Apraxia
Keywords: apraxia; occupational therapy; multiple sclerosis; manual dexterity
MeSH Terms: conditions — Multiple Sclerosis; Apraxias | interventions — Occupational Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Occupational therapy using a special arm function training.
  Interventions: Other: Occupational Therapy
- Group 2 (Active Comparator): Physical therapy using the Theraband for training of force.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Occupational Therapy — Occupational therapy using a special arm function training.
  Arms: Group 1
Other: Physical therapy — Physical therapy for arm force training.
  Arms: Group 2

SUMMARY:
Limb apraxia is defined as the inability to correctly perform skilled and/or learned limb movements, which cannot be explained by elementary motor and sensory deficits or cognitive problems. Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system and the leading cause of disability in young adults. Apraxia and impaired manual dexterity are common problems in patients with MS leading to impaired activities of daily living. However, a specific training program to improve apraxia as well as manual dexterity in MS is lacking.

In this study, the investigators want to evaluate the impact of a targeted occupational therapy program on apraxia and manual dexterity in patients with MS that have dexterity problems.

Patients routinely seen in the investigators MS consulting hour, fulfilling all inclusion and exclusion criteria and willing to participate in the study will be evaluated for Apraxia and manual dexterity. In case of Apraxia and/or impaired manual dexterity, patients will be randomized 1:1 using sealed envelopes to receive occupational home therapy (experimental group) or general physical exercises (control group) for 4 weeks.

At study entry and study end after 4 weeks, apraxia and manual dexterity will be tested in all patients.

DETAILED DESCRIPTION:
Background

Limb apraxia is defined as the inability to correctly perform skilled and/or learned limb movements, which cannot be explained by elementary motor and sensory deficits or cognitive problems. It impairs real object/tool use as well as pantomime and imitation of gestures affecting both sides of the body and can be a major source of disability independent of other neurological deficits. It significantly affects activities of daily living (ADL) and is associated with poorer outcome for independent living or return to work.

Apraxia is largely based on left parieto-frontal damage due to focal injury or more widespread neurodegeneration of cortical areas and/or their connections. However, apraxia has been described in damage of the right hemisphere, although less frequent and severe.

Apraxia is increasingly recognized as a clinical problem in restorative neurology and various approaches were described how to treat the disorder.

Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system and the leading cause of disability in young adults. It is characterized by focal demyelination as well as axonal damage. MS has been classically thought of as a typical white matter disorder. However, early pathology studies and recent magnetic resonance tomography (MRI) studies show demyelination in the cortex and deep gray matter nuclei. Grey matter damage starts early in the disease and substantially affects cognitive functioning.

Apraxia and impaired manual dexterity are common problems in MS leading to impaired activities of daily living. However, a specific training program to improve apraxia and manual dexterity in MS is lacking. In this study, we want to evaluate the impact of a targeted occupational therapy program on apraxia and manual dexterity in patients with MS that have dexterity problems.

It is a rater-blind, randomized, controlled trial. Patients routinely seen in our MS consulting hour, fulfilling all inclusion and exclusion criteria and willing to participate in the study will be evaluated for Apraxia using the AST (Apraxia Screen of TULIA). In case of Apraxia patients will be randomized 1:1 using sealed envelopes to receive occupational home therapy (experimental group) or general physical exercises (control group) for 4 weeks (4 times 5 days in a row).

At study entry and study end after 4 weeks, apraxia will be tested in all patients using the extended version of the AST, the TULIA. Furthermore, a questionnaire on "activities of daily living" and "quality of life" will be evaluated, and test regarding cognition, spasticity, ataxia, fatigue as well as the EDSS will be performed.

Objective

To evaluate the impact of a targeted occupational therapy program on apraxia and manual dexterity in patients with MS.

Methods

see above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with all forms of MS
* Age 18-60 years

Exclusion Criteria

* Any disease other than multiple sclerosis that could possibly explain the patient's signs and symptoms
* A relapse which started within 60 days prior to the examination
* Uncontrolled, clinically significant heart diseases, such as arrhythmias, angina, Coronary heart disease or uncompensated congestive heart failure, medication with glycosides.
* A history of drug abuse in the 6 months prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in apraxia score as measured by TULIA | From day of randomisation to end of study, expected to be after 4 weeks

SECONDARY OUTCOMES:
Change in manual dexterity | From day of randomisation to end of study, expected to be after 4 weeks
  Measured by the coin rotation task and 9-hole-peg-test
Change in activities of daily living | From day of randomisation to end of study, expected to be after 4 weeks
  Measured by questionnaire
Change in quality of life | From day of randomisation to end of study, expected to be after 4 weeks
  Measured by questionnaire
Change in fatigue | From day of randomisation to end of study, expected to be after 4 weeks
  Measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Kamm, MD, Principal Investigator — Department of Neurology, Inselspital Bern, 3010 Bern, Switzerland
Locations (1):
- Department of Neurology, Bern university Hospital, Bern, Switzerland

REFERENCES:
- [Background] Vanbellingen T, Kersten B, Van de Winckel A, Bellion M, Baronti F, Muri R, Bohlhalter S. A new bedside test of gestures in stroke: the apraxia screen of TULIA (AST). J Neurol Neurosurg Psychiatry. 2011 Apr;82(4):389-92. doi: 10.1136/jnnp.2010.213371. Epub 2010 Oct 9. PMID 20935324
- [Background] Bohlhalter S, Vanbellingen T, Bertschi M, Wurtz P, Cazzoli D, Nyffeler T, Hess CW, Muri R. Interference with gesture production by theta burst stimulation over left inferior frontal cortex. Clin Neurophysiol. 2011 Jun;122(6):1197-202. doi: 10.1016/j.clinph.2010.11.008. Epub 2010 Dec 3. PMID 21130031
- [Derived] Kamm CP, Mattle HP, Muri RM, Heldner MR, Blatter V, Bartlome S, Luthy J, Imboden D, Pedrazzini G, Bohlhalter S, Hilfiker R, Vanbellingen T. Home-based training to improve manual dexterity in patients with multiple sclerosis: A randomized controlled trial. Mult Scler. 2015 Oct;21(12):1546-56. doi: 10.1177/1352458514565959. Epub 2015 Jan 26. PMID 25623246